CLINICAL TRIAL: NCT00142168
Title: Phase II Study of CC-5103 and Rituximab in Waldenstrom's Macroglobulinemia
Brief Title: CC-5013 (Lenalidomide) and Rituximab in Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxicity
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-158
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: CC-5103 (lenalidomide); rituximab; Waldenstrom's macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-5103 (Lenalidomide) and Rituximab (Experimental): Intended therapy consisted of 48 weeks of CC-5103 (lenalidomide)(25 mg/d for 3 weeks and then 1 week off) along with rituximab (375 mg/m(2)/wk) dosed on weeks 2 to 5 and 13 to 16.
  Interventions: Drug: CC-5103 (lenalidomide); Drug: Rituximab

INTERVENTIONS:
Drug: CC-5103 (lenalidomide) — Taken orally once a day for 21 days followed by 7 days of no CC-5103 (lenalidomide)
  Other Names: lenalidomide; Revlimid
Drug: Rituximab — Begins on week 2 of treatment and is given intravenously once a week for 4 weeks
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the number of patients with Waldenstrom's macroglobulinemia that will benefit from treatment with CC-5103 (lenalidomide) and rituximab, what the side effects are and how long the benefit will last.

DETAILED DESCRIPTION:
* The study drug CC-5103 (lenalidomide) will be administered orally once daily for 21 days followed by 7 days of no CC-5103 (lenalidomide) (this will be one 28 day treatment cycle). This cycle will repeat itself every 28 days as long as the patient is tolerating the medication and there is no disease progression.
* Starting on the second week, patients will begin treatment with rituximab intravenously once a week for 4 weeks (week 2-5). Prior to each treatment, patients will receive medications to prevent or reduce the side effects of rituximab (benadryl, tylenol and possible decadron). During the infusion, the patients' blood pressure and pulse will be monitored frequently and the rate of infusion may decrease depending upon the side effects. Blood work will also be performed each week.
* On week 12 the disease status will be evaluated. A physical exam, blood test, CT scan and bone marrow biopsy may be repeated if necessary to fully evaluate the disease. If the disease has gone away completely, some tests may be repeated again to confirm this.
* If the disease has gotten worse after 12 weeks, then the patient will be removed from the study.
* If the disease is stable or getting better, the patient will continue with therapy. During weeks 13-16 rituximab infusions will be repeated and CC-5103 will continue to be taken daily for 21 days followed by 7 days of rest. This 28 day cycle may be repeated until the patient has completed 48 weeks (12 months) of treatment as long as the side effects are acceptable and the disease does not progress.
* All patients will undergo an off-study evaluation that includes a physical exam, blood work, CT scans and bone marrow biopsy. If the patient completes 78 weeks of therapy and the disease does not get worse, they will be evaluated every 12 weeks to determine the status of their disease for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia using consensus panel criteria
* Age 18 years or older
* CD20 positive based on any previous bone marrow immunohistochemistry or flow cytometric analysis
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study
* Measurable disease, defined as presence of immunoglobulin M paraprotein with a minimum IgM level of equal to or greater than 2 times the upper limit of normal.
* ECOG performance status of 0-2
* Absolute neutrophil count ≥ 100,000,000/L
* Platelet count ≥ 50,000,000,000/L
* Hemoglobin > 8 g/dL
* Serum creatinine < 2.5 mg/dL
* Total bilirubin < 1.5 mg/dL
* AST and ALT < 2.5 x ULN
* Disease free of prior malignancies fir 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness
* Pregnant or lactating women
* Prior therapy with rituximab or CC-5103
* Known hypersensitivity to thalidomide
* Development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Concurrent use of other anti-cancer agents or treatments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Insitute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Result] Treon SP, Soumerai JD, Branagan AR, Hunter ZR, Patterson CJ, Ioakimidis L, Chu L, Musto P, Baron AD, Nunnink JC, Kash JJ, Terjanian TO, Hyman PM, Nawfel EL, Sharon DJ, Munshi NC, Anderson KC. Lenalidomide and rituximab in Waldenstrom's macroglobulinemia. Clin Cancer Res. 2009 Jan 1;15(1):355-60. doi: 10.1158/1078-0432.CCR-08-0862. PMID 19118065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient clinic at DFCI
Pre-assignment Details: Symptomatic WM patients requiring therapy
Groups:
- Lenalidomide and Rituximab: Intended therapy consisted of 48 weeks of lenalidomide (25 mg/d for 3 weeks and then 1 week off) along with rituximab (375 mg/m(2)/wk) dosed on weeks 2 to 5 and 13 to 16.
Period: Overall Study
Arm/Group | Lenalidomide and Rituximab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression is measured as the length in time in months from starting therapy until progression, defined as 25% increase in serum IgM from nadir.
Time Frame: 34.3 months
Population: All enrolled patients
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 16
months | 17.1 [2 to 34.3]

2. Primary Outcome: Overall Response
Description: Overall response is the total number of participants who respond to therapy. Patients achieving a complete response (CR) will be defined as having achieved resolution of all symptoms, normalization of their serum IgM levels with complete disappearance of their IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly during any point while in this study and normal bone marrow biopsy. Patients achieving a partial response (PR) and a minor response (MR) will be defined as achieving a > 50% and > 25% reduction in serum IgM levels, respectively, during any point while in this study. Patients with stable disease (SD) will be defined as having < 25% change in serum IgM levels, in the absence of new or increasing adenopathy or splenomegaly and/or other progressive signs or symptoms of WMduring any point while in this study.
Time Frame: 34.3 months
Population: Evaluable patients. 4 participants were withdrawn for adverse events and were unevaluable.
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 12
participants | 8

3. Secondary Outcome: Major Response Rate
Description: Major response rate is the number of participants who achieve at a PR or better. A PR or better will be defined as achieving a >50% reduction in serum IgM levels.
Time Frame: 34.3 months
Population: Evaluable patients. 4 participants were withdrawn for adverse events and were unevaluable.
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 12
participants | 4

4. Secondary Outcome: Minor Response Rate
Description: A minor response is defined as having achieved >25% but less than 50% reduction in serum IgM levels.
Time Frame: 34.3 months
Population: Evaluable patients. 4 participants were withdrawn for adverse events and were unevaluable.
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Rituximab
Number analyzed (Participants) | 12
participants | 4

ADVERSE EVENTS:
Arm/Group | Lenalidomide and Rituximab
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 8/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Rituximab (N=16)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) — 5 patients developed grade 3 neutropenia
Anemia (Blood and lymphatic system disorders) | 1 (1) — 1 patient, grade 3
arrythmia (Cardiac disorders) | 1 (1) — 1 patient, grade 3
chest pain (Cardiac disorders) | 1 (1) — 1 patient, grade 3
pulmonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 patient, grade 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — 1 patient, grade 3
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 patient, grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide and Rituximab (N=16)
Anemia (Blood and lymphatic system disorders) | 8 (8) — 1 patient grade 3

LIMITATIONS AND CAVEATS:
Due to toxicity, study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No